CLINICAL TRIAL: NCT00285519
Title: The Effects of Controlling Morning Hypertension on Target Organ Damage With Adrenergic Blockers, Based on Self-Measured Morning Blood Pressure Readings
Brief Title: Japan Morning Surge-1 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Japan Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHF-03-143
Record Dates: First submitted 2006-01-24; First posted 2006-02-02 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2006-02

CONDITIONS: Hypertension
Keywords: Morning hypertension
MeSH Terms: conditions — Hypertension | interventions — Doxazosin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Doxazosin (drug)

SUMMARY:
The purpose of this study is to examine whether strict blood pressure (BP) control by doxazosin using home BP monitoring, especially targeting the morning BP level, can reduce hypertensive target organ damage.

DETAILED DESCRIPTION:
Morning blood pressure may play an important role in the pathogenesis of hypertensive target organ damage. Increased sympathetic nerve activity is reported to be one of the mechanisms of morning hypertension; however, there are no available data that show whether strict home blood pressure control, especially in the morning period, can reduce target organ damage.We will evaluate whether strict morning blood pressure control by sympathetic nervous system blockade using an alfa-blocker, doxazosin, and with the addition of a beta-blocker if needed, can reduce hypertensive target organ damage.

ELIGIBILITY:
Inclusion Criteria:

* Morning systolic blood pressure >135 mmHg in a sitting position at home while on stable antihypertensive medication for at least 3 months

Exclusion Criteria:

* History of heart failure
* Presence of orthostatic hypotension, dementia, malignancy and chronic inflammatory disease
* Taking an alfa-blocker or beta-blocker
* Atrial fibrillation or atrial flutter

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2003-08; Study Completion 2005-08

PRIMARY OUTCOMES:
brain natriuretic peptide and the urinary albumin excretion/creatinine ratio at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, MD, PhD, Study Chair — Division of Cardiovascular Medicine, Department of Medicine, Jichi Medical University School of Medicine
Locations (1):
- Division of Cardiovascular Medicine, Department of Medicine, Jichi Medical University School of Medicine, Shimotsuke, Tochigi, Japan

REFERENCES:
- [Derived] Hoshide S, Parati G, Matsui Y, Shibazaki S, Eguchi K, Kario K. Orthostatic hypertension: home blood pressure monitoring for detection and assessment of treatment with doxazosin. Hypertens Res. 2012 Jan;35(1):100-6. doi: 10.1038/hr.2011.156. Epub 2011 Sep 15. PMID 21918522